CLINICAL TRIAL: NCT07087899
Title: Romatoid Artritli Hastalarda Müziğin Semptom Yönetimi ve Yaşam Kalitesi Üzerine Etkisi
Brief Title: The Effect of Music on Symptom Management and Quality of Life in Patients withRheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Irem Yildiz Cilengiroglu (Other)
Collaborators: Trakya University (Other)
Responsible Party: Sponsor-Investigator, Irem Yildiz Cilengiroglu, Research assistant, Trakya University
Organization: Trakya University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2023/73
Record Dates: First submitted 2025-07-03; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Rheumatoid Arthritis; Music; Symptoms Arthritis
Keywords: rheumatoid arthritis; music; quality of life; symptom management
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- music (Experimental): The participants were informed about the research process during the first meeting. Participants were told that, if they agreed to participate in the study, they would need to listen to music twice a day-once during the day and once at night-for a period of one month. It was explained that each participant would be provided with a music player and headphones for one month, and that these items would need to be returned after the study ended. Participants were also given information on how to listen to the music. Participants were instructed on how to use the music player, informed that there were two playlists-one for daytime and one for nighttime-and advised to listen to each playlist for a maximum of 30 minutes.
  Interventions: Other: music
- control (No Intervention): In the first interview, participants were informed about the research process. Patient information forms and scales (EQ-5D General Quality of Life Scale, DAS-28 Disease Activity Score and Patient Symptom Thermometer) that would be used in data collection were explained to the participants. Participants were informed about how often and how these forms and scales would be applied. No intervention was applied to the participants in the control group in the study.

INTERVENTIONS:
Other: music — listening music
  Arms: music

SUMMARY:
This randomized controlled study was designed to determine the effects of music on symptom management and quality of life in patients with rheumatoid arthritis.

The study was conducted between October 2023 and August 2024 with 88 patients diagnosed with rheumatoid arthritis (41 experimental, 47 control) at the Rheumatology clinic and outpatient clinic of a university hospital in Edirne. Within the scope of this study, the Turkish validity and reliability of the Patient Symptom Thermometer scale were tested. Data were collected using the "Patient Information Form" including sociodemographic and disease-related characteristics, the "EQ-5D General Quality of Life Scale," the "Patient Symptom Thermometer," and the "DAS-28 Disease Activity Score."

DETAILED DESCRIPTION:
Background and Aim: Rheumatoid arthritis is a chronic disease that significantly reduces quality of life due to both physical and psychosocial symptoms. Complementary methods such as music therapy are thought to be effective in alleviating symptoms and improving quality of life in patients with rheumatoid arthritis. This randomized controlled study was designed to determine the effects of music on symptom management and quality of life in patients with rheumatoid arthritis.

Material and Methods: The study was conducted between October 2023 and August 2024 with 88 patients diagnosed with rheumatoid arthritis (41 experimental, 47 control) at the Rheumatology clinic and outpatient clinic of a university hospital in Edirne. Within the scope of this study, the Turkish validity and reliability of the Patient Symptom Thermometer scale were tested. Data were collected using the "Patient Information Form" including sociodemographic and disease-related characteristics, the "EQ-5D General Quality of Life Scale," the "Patient Symptom Thermometer," and the "DAS-28 Disease Activity Score." During the first interview, the relevant scales and questionnaire were applied to patients in both the experimental and control groups. Patients in the experimental group were provided with music players and headphones to listen to music twice a day-once during the day and once at night-for one month. On the 15th and 30th days of the study, the EQ-5D General Quality of Life Scale and the Patient Symptom Thermometer were administered to the experimental group. The same scales were also applied to the control group, who did not listen to music, on the 15th and 30th days.

Financial Support: The present study was supported by the Research Fund of Trakya University. Project No: 2023/73

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with RA by a physician according to the American College of Rheumatology - The European Alliance of Associations for Rheumatology (ACR-EULAR) 2010 criteria
* Patients diagnosed with Rheumatoid Arthritis at least 6 months ago
* Patients with Rheumatoid Arthritis who volunteer to participate in the study

Exclusion Criteria:

* Patients with hearing problems
* Rheumatoid Arthritis patients who do not volunteer to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2023-12-23 (Actual); Study Completion 2024-08-25 (Actual)

PRIMARY OUTCOMES:
quality of life score | one month
  Change in the mean scores of the EQ-5D General Quality of Life Scale of the patients at the first interview, on the 15th day and on the 30th day
Patient Symptom Thermometer scores | one month
  Change in mean Patient Symptom Thermometer scores of patients at the first visit, on the 15th day, and on the 30th day

CONTACTS AND LOCATIONS:
Overall Officials: Yıldız Çilengiroğlu, Principal Investigator — Trakya University
Locations (1):
- Trakya University, Edirne, Turkey (Türkiye)